CLINICAL TRIAL: NCT07086196
Title: Retrospective Analysis of Real-World Outcomes of Ribociclib in First-Line Treatment for Metastatic HR+/HER2- Breast Cancer
Brief Title: A Study of Real-World Outcomes of Ribociclib in First-Line Treatment for Metastatic HR+/HER2- Breast Cancer
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011AUS72
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Metastatic HR+/HER2- Breast Cancer
Keywords: Hormone receptor; Human epidermal growth factor receptor 2; Breast cancer; Administrative claims
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Ribociclib Cohort: Patients who received ribociclib as 1L treatment for HR+/HER2- mBC.

SUMMARY:
The main aim of this study was to describe the profile of hormone receptor positive/human epidermal growth factor receptor 2 negative (HR+/HER2-) metastatic breast cancer (mBC) patients who received first-line (1L) current treatment options with ribociclib in the United States (US) clinical practice.

This study used administrative claims data. De-identified patient-level data of adult patients with HR+/HER2- mBC who initiated 1L treatment with a cyclin dependant kinase 4/6 inhibitor (CDK4/6i) i.e., ribociclib from the Komodo Health Solutions Research Database (KRD; data from 1 January 2016 to 30 June 2023) was used. Data included medical and pharmacy claims for insured patients, which had already been collected (i.e., secondary use of data).

ELIGIBILITY:
Inclusion criteria:

* Had 1 or more paid pharmacy claims for ribociclib with the first claim for the CDK4/6i observed between 26 February 2018 and 31 December 2022 (i.e., during the index period)

  * With the index CDK4/6i used in combination with an endocrine-based therapy, that is an aromatase inhibitor (i.e., letrozole, anastrozole, or exemestane), or fulvestrant, as 1L treatment for mBC
  * With the endocrine therapy (ET) initiated within 60 days of the first paid pharmacy claim of the index CDK4/6i; ET may have been initiated no earlier than 60 days prior to the index date (expected window for insurance approval of the CDK4/6i as 1L treatment for mBC in a real-world setting)
* Adult who was 18 years of age or older as of the index date
* Had 2 or more medical service claims with a code for breast cancer (BC) separated by 30 days or more, and 1 or more claims with a code for BC prior to the index date
* Had 2 or more medical service claims with a code for a secondary neoplasm separated by 30 days or more, with the first code for a secondary neoplasm occurring not earlier than 30 days from the first diagnosis for BC, and 1 or more claims with a code for a secondary neoplasm prior to the index date
* Had continuous health plan enrollment for 12 months or more prior to and 1 month or more after the index date

Exclusion criteria:

* Patients who did not meet the inclusion criteria
* Had a diagnosis for other primary cancers (other than BC) before the first diagnosis for secondary neoplasm
* Had prior treatments for BC (i.e., chemotherapy, targeted therapy, ET [except ≤60 days prior to index date], or immunotherapy) during the 12-month washout period (relapsed/progressed ≤12 months prior to index date)
* Had prior surgical procedure for BC during the 12-month washout period (relapsed/progressed ≤12 months prior to index date)
* Had evidence of participation in a clinical trial prior to or at the index date (International Classification of Disease, 10th Edition, Clinical Modification [ICD-10-CM]: Z00.6)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, non-interventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Number Patients by Demographic Category | Baseline
  Demographics included:
  * Age (≥ 65 years, ≥ 75 years)
  * Gender
  * Race
  * Index year (year of the first paid pharmacy claim for ribociclib)
Number of Patients by Clinical Characteristic Category | Baseline
  Clinical characteristic categories included:
  * Menopausal status
  * Comorbidity
  * Metastatic site
  * Eastern Cooperative Oncology Group (ECOG) performance score less than 2
  ECOG performance score measures a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability. Scores range from 0 (fully active, able to carry out all pre-disease performance without restriction) to 5 (deceased).
Clinical Characteristic: National Cancer Institute (NCI) Comorbidity Index Score | Baseline
  The NCI comorbidity index is a tool used to measure the risk of non-cancer deaths for cancer patients based on the presence and severity of other health conditions. It includes 14 conditions identified using administrative data diagnosis and procedure codes. The index excludes solid tumors, leukemias, and lymphomas as comorbid conditions. Each condition is assigned a score based on how serious it is and patient scores are summed to give a final overall score. A high score indicates a higher burden of comorbid conditions and possible higher risk of death.
Clinical Characteristic: Number of Metastatic Sites | Baseline
Treatment Characteristic: Number of Patients by Type of Treatment Received While on 1L mBC Treatment | Up to approximately 3 years and 4 months
  Treatments included:
  * Endocrine therapy partner (AI, Fulvestrant, or AI and Fulvestrant)
  * Gonadotropin-releasing hormone (GNRH)
  * Cytochrome P450, family 3, subfamily A (CYP3A) inhibitors and inducers
  * P-inhibitors and inducers
  * Medications potentially associated with an increased risk of torsade de pointes
Treatment Characteristic: Time from mBC diagnosis to 1L Initiation | Baseline
Treatment Characteristic: Duration of Follow-up From 1L Initiation | Up to approximately 3 years and 4 months
Treatment Characteristic: Duration of 1L mBC Treatment | Up to approximately 3 years and 4 months

SECONDARY OUTCOMES:
Number of Patients by Tolerability-related Medical Events Experienced While on 1L Treatment With Ribociclib | Up to approximately 3 years and 4 months
  Medical events were assessed among patients who did not have the selected condition during the baseline period and were described based on the presence of 2 or more medical claims on distinct dates.
Number of Patients by Cardiovascular-related Medical Events Experienced While on 1L Treatment With Ribociclib | Up to approximately 3 years and 4 months
  Medical events were assessed among patients who did not have the selected condition during the baseline period and were described based on the presence of 2 or more medical claims on distinct dates.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States